CLINICAL TRIAL: NCT00758693
Title: Frontline Treatment With Bendamustine in Combination With Rituximab in Adults Age 65 or Older With Chronic Lymphocytic Leukemia: A Phase II Study
Brief Title: Frontline Treatment With Bendamustine in Combination With Rituximab in Adults Age 65 or Older With Chronic Lymphocytic Leukemia (CLL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn due to insufficient accrual
Sponsor: University of Kentucky (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-LEUK-07-MCC/CI
Record Dates: First submitted 2008-09-19; First posted 2008-09-25 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Bendamustine; Treanda; Rituximab; Rituxan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Bendamustine + Rituximab
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine 100 mg/m2 intravenously on days 1 and 2 on a 28-day cycle for 6 cycles
  Other Names: Treanda
Drug: Rituximab — Rituximab 500 mg/m2 on a 28-day cycle for 6 cycles
  Other Names: Rituxan

SUMMARY:
Many chemotherapy combinations may be used to treat patients with chronic lymphocytic leukemia (CLL). Although there are many options, a single, best option is not agreed upon by most cancer specialists. Bendamustine, a medicine recently approved for use in the United States, has been used in combination with rituximab in previous studies to treat patients whose CLL has returned after previous standard treatments. The purpose of this study is to determine whether bendamustine with rituximab is effective for the initial treatment of CLL for patients aged 65 and older.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed chronic lymphocytic leukemia.
* A minimum of any one of the following disease-related symptoms must be present:

  * Weight loss ≥10% within the previous 6 months.
  * Extreme fatigue (ie, ECOG PS 2; cannot work or unable to perform usual activities).
  * Fevers of greater than 100.5"F for ≥ 2 weeks without evidence of infection.
  * Night sweats without evidence of infection. or
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia or
  * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy or
  * Massive (ie, >6 cm below the left costal margin) or progressive splenomegaly or
  * Massive nodes or clusters (ie, > 10 cm in longest diameter) or progressive lymphadenopathy or
  * Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months but
  * Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for protocol therapy
* No prior therapy for CLL is allowed. Participants may have taken corticosteroids previously but must be ≥ 28 days from last dose prior to enrolment.
* Age >65 years.
* Life expectancy of greater than 1 year.
* ECOG performance status better than or equal 2.
* Patients must have normal organ and marrow function as defined below:

  * total bilirubin within normal institutional limits unless resulting from documented hemolysis
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had previous chemotherapy or radiotherapy for the treatment of CLL.
* Patients may not be receiving any other investigational agents.
* Patients with known brain involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bendamustine or rituximab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with a known history of viral hepatitis, with the exception of Hepatitis A that has recovered.
* Patients who require concomitant treatment with CYP1A2 inhibitors including: Cimetidine, Ciprofloxacin, Fluvoxamine, Ticlopidine.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the response rate | Defined by the 1996 NCI sponsored working group guidelines for the diagnosis and treatment of CLL

SECONDARY OUTCOMES:
Describe the toxicity rates and severities | Up to 2 years after enrollment
Describe the quality of life participants experience while receiving this combination therapy | Up to 2 years after enrollment
Determine the health utility scores of participants while receiving this combination therapy | Up to 2 years after enrollment
Conduct exploratory analyses of associations between clinical responses and protein expression and phosphorylation using novel flow cytometry methods | Pre and Post treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Hayslip, MD, MSCR, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- See also: Markey Cancer Center Blood and Marrow Transplant Study Search — http://markey.uky.edu/studysearch/default.aspx?site=Blood%20and%20Marrow%20Transplant